CLINICAL TRIAL: NCT03880539
Title: Historically-controlled Clinical Trial of the Efficacy and Safety of Bezlotoxumab (BEZLO) in Addition to Standard of Care (SOC) Vancomycin for the Treatment of Multi-recurrent Clostridium Difficile Infection (CDI)
Brief Title: Bezlotoxumab (BEZLO) In Addition To Standard Of Care (SOC) Vancomycin For The Treatment of Multi-Recurrent Clostridium Difficile Infection
Acronym: BEZLO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Lisa Clough, Principal Investigator, University of Kansas Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Study00143405
Record Dates: First submitted 2019-03-11; First posted 2019-03-19 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Clostridium Difficile Infection Recurrence
Keywords: C.diff; Clostridium Difficile; recurrence; Bezlotoxumab; CDI
MeSH Terms: conditions — Recurrence | interventions — bezlotoxumab; Vancomycin

STUDY DESIGN:
Intervention Model Description: The intervention group will consist of a single arm of patients treated with BEZLO + SOC oral VAN pulse/taper for multi-recurrent CDI, with a planned enrollment of 12 patients. To achieve the aim of the proposed study, we will compare the efficacy of BEZLO + SOC oral VAN pulse/taper to a historical cohort of patients treated with SOC oral VAN pulse/taper only. These patients will be matched 1:6 on criteria previously outlined in this proposal (BEZLO + SOC, n=12; SOC comparator, n=72; total number of patients in study, n=84).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- BEZLO + SOC taper (Other): Single arm of patients treated with BEZLO + SOC oral VAN pulse/taper.
  Interventions: Drug: bezlotoxumab; Drug: Vancomycin Oral

INTERVENTIONS:
Drug: bezlotoxumab — Adding BEZLO to SOC oral VAN pulse/taper
  Other Names: Zinplava
Drug: Vancomycin Oral — SOC vancomycin pulse/taper
  Other Names: Firvanq

SUMMARY:
This is a research study to collect information from people that have Clostridium difficile infection (CDI) and are treated with a standard antibiotic treatment in which the antibiotic dose is gradually reduced over 6 weeks and bezlotoxumab (BEZLO), an approved monoclonal antibody targeting C. difficile toxin, which has shown to reduce CID recurrence when used in combination with standard antibiotic treatment.

DETAILED DESCRIPTION:
Clostridium difficile (C. diff) is a type of bacteria which causes diarrhea in some people who receive antibiotics for other infections. The current antibiotics used to treat C diff infection (CDI) are usually successful in treating the initial episode of CDI, but may not prevent recurrent infection. To prevent recurrent CDI, standard oral antibiotic treatment with vancomycin is extended by gradually reducing the dose over 4-8 weeks. This is called antibiotic taper. Bezlotoxumab (BEZLO), a monoclonal antibody targeting C. difficile toxin B, is an approved medication that has also been shown to reduce CDI recurrence in patients receiving antibacterial drug treatment of CDI. In this study, approximately 12 people with multi-recurrent CDI will be treated with BEZLO in combination with standard oral tapered vancomycin. Study participation will last 16 weeks. The rate of CDI recurrence in this group will be compared to information collected from approximately 72 historical patients with multi-recurrent CDI treated with oral tapered vancomycin only.

ELIGIBILITY:
Inclusion Criteria (Interventional):

* i) age 18 years or older;
* ii) diagnosis of multi-recurrent CDI, defined as passage of 3 or more loose stools in 24 hours or less for at least 2 consecutive days and a positive stool test for toxigenic C. difficile (nucleic acid amplification test [NAAT] and toxin enzyme immunoassay [EIA] positive), with 2 or more confirmed prior CDI episodes;
* iii) receiving or planning to receive a 10- to 14-day course of SOC therapy with oral VAN followed by a tapered VAN regimen for at least 4 weeks;
* iv) patient highly unlikely to become pregnant due to being female and not of reproductive potential or female of reproductive potential agreeing to be abstinent or using 2 acceptable methods of birth control starting at enrollment and through the 16-week study period; and
* v) patient or legal representative voluntarily agreeing to participate by providing written informed consent after the nature of the study has been fully explained.

Inclusion Criteria (Historical Control):

* i) age 18 years or older
* ii) diagnosis of multi-recurrent CDI
* iii) received 10- to 14-day course of SOC therapy with oral VAN followed by a tapered VAN regimen.

Exclusion Criteria:

* i) active chronic diarrheal illness, such as (but not limited to) ulcerative colitis or Crohn's disease or with a condition such that they routinely pass loose stool
* ii) planned surgery for CDI within 24 hours
* iii) positive pregnancy test in the 48 hours before the infusion or unwilling to undergo pregnancy testing if a pre-menopausal female who is not sterilized and therefore has the potential to bear a child
* iv) breastfeeding or planning to breastfeed prior to the completion of the study period
* v) previous receipt of BEZLO
* vi) receipt of immune globulin within 6 months prior to enrollment or planning to receive immune globulin prior to completion of the 16-week study period
* vii) receipt of non-SOC CDI therapy within 14 days prior to enrollment
* viii) planned treatment with SOC therapy for longer than 6 weeks
* ix) receipt of medications to control diarrhea such as loperamide, diphenoxylate hydrochloride/atropine sulfate at any time prior to completion of the 16-week study period
* x) medical history of decompensated congestive heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2021-11-18 (Actual)

PRIMARY OUTCOMES:
Rate of CDI reoccurrence at 12 weeks | 12 weeks
  If diarrhea resolves (defined as <2 loose stools per day for at least 2 consecutive days) and subsequently begins again (3 or more loose stools in 24 hours or less for at least 2 consecutive days), this will represent a new episode of diarrhea. If there is a new episode of diarrhea at any time during the 12-week study period, an unscheduled visit will be conducted. A stool sample will be provided for any new episode of diarrhea which occurs and a stool test for toxigenic C. difficile (NAAT plus EIA) will be performed. CDI reoccurrence will be defined as new episode of diarrhea and positive stool test for toxigenic C. difficile (NAAT plus EIA).

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A Clough, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States